CLINICAL TRIAL: NCT03527550
Title: A Randomized Controlled Trial of Cognitive Control Training for Urgency in a Naturalistic Clinical Setting
Brief Title: Cognitive Control Training for Urgency in a Naturalistic Clinical Setting
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data collection ended due to COVID-19 (study site closed to in-person visits)
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrew D. Peckham, Research Fellow, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2017P001550; 1F32MH115530 (NIH)
Record Dates: First submitted 2018-04-19; First posted 2018-05-17 (Actual); Results first posted 2021-03-25 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Impulsive Behavior; Mental Disorders
Keywords: impulsivity; Inhibition (Psychology); Working memory; Cognitive Remediation
MeSH Terms: conditions — Impulsive Behavior; Mental Disorders; Inhibition, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training plus Treatment as Usual (Experimental): Participants in this arm will receive daily computerized cognitive training sessions during partial hospitalization, in addition to treatment as usual. Cognitive training sessions will alternate between response inhibition training and working memory training.
  Interventions: Other: Cognitive Control Training
- Treatment as Usual (TAU) (No Intervention): Participants in the Treatment As Usual group will receive usual treatment in the partial hospitalization program.

INTERVENTIONS:
Other: Cognitive Control Training — Cognitive Control Training involves daily practice with one of two computerized interventions. The first intervention is an adaptive Go/No-Go task to provide practice in the domain of response inhibition. Participants press a key as fast as possible in response to stimuli (letters of the alphabet), but must inhibit responses to a specific letter. The second intervention is an adaptive Paced Auditory Serial Addition Task (PASAT), designed to practice working memory. Participants are presented with single numbers presented aurally, and must add each number they hear to the previous number and click the correct sum on the screen.
  Arms: Cognitive Training plus Treatment as Usual

SUMMARY:
This study is designed to test whether computer-based cognitive exercises are helpful for reducing a specific type of impulsivity. Also, the study is testing whether these are exercises are associated with specific changes in behavior and in the brain. Participants will be psychiatric patients enrolled in a partial hospitalization program. Half of these participants will receive usual treatment, and half will complete computer-based cognitive exercises in addition to usual treatment.

DETAILED DESCRIPTION:
Impulsivity has different components. One personality trait related to impulsivity, known as "urgency," is strongly related to many different mental health symptoms and risky behaviors. Urgency refers to impulsivity specifically in the context of strong emotions.

Research shows that higher levels of urgency are related to specific deficits in cognition. Problems with response inhibition--the ability to cancel or withhold a planned action--are associated with urgency. Also, research shows that difficulties in another aspect of cognition--working memory--may moderate the relationship between inhibition deficits and urgency. One previous study found that people who practiced computerized response inhibition and working memory tasks for two weeks reported significant decreases in urgency.

It is unknown if these computerized tasks would be helpful for reducing urgency in adults with psychiatric disorders. Furthermore, it is unknown if changes in urgency are related to changes in the brain mechanisms that help to support response inhibition. This study will collect data on brain activity while people are completing response inhibition tasks.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving treatment at the McLean Hospital Behavioral Health Partial Hospital Program (PHP)
* Report an average score of 3.0 or greater on the Negative Urgency scale, the Positive Urgency scale, or 3.0 or greater on both scales, upon admission to the PHP
* Right-handed (if enrolled in EEG arm)

Exclusion Criteria:

* Currently undergoing electroconvulsive therapy (ECT)
* Current symptoms of acute mania
* Current symptoms of acute psychosis
* History of traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of data analysis, de-identified data from this study will be made available to the National Database for Clinical Trials Related to Mental Illness (NDCT).
Supporting Information: Study Protocol
Time Frame: Data will be made available when primary data analysis is complete.
Access Criteria: Data will be made available to users of the NDCT website:
  https://data-archive.nimh.nih.gov/
URL: https://data-archive.nimh.nih.gov/

REFERENCES:
- [Background] Peckham AD, Johnson SL. Cognitive control training for emotion-related impulsivity. Behav Res Ther. 2018 Jun;105:17-26. doi: 10.1016/j.brat.2018.03.009. Epub 2018 Mar 27. PMID 29609103
- [Derived] Peckham AD, Sandler JP, Dattolico D, McHugh RK, Johnson DS, Bjorgvinsson T, Pizzagalli DA, Beard C. Cognitive control training for urgency: A pilot randomized controlled trial in an acute clinical sample. Behav Res Ther. 2021 Nov;146:103968. doi: 10.1016/j.brat.2021.103968. Epub 2021 Sep 14. PMID 34562728

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive Training Plus Treatment as Usual: Participants in this arm received daily computerized cognitive training sessions during partial hospitalization, in addition to treatment as usual. Cognitive training sessions alternated between response inhibition training and working memory training.
  Cognitive Control Training: Cognitive Control Training involves daily practice with one of two computerized interventions. The first intervention is an adaptive Go/No-Go task to provide practice in the domain of response inhibition. Participants press a key as fast as possible in response to stimuli (letters of the alphabet), but must inhibit responses to a specific letter. The second intervention is an adaptive Paced Auditory Serial Addition Task (PASAT), designed to practice working memory. Participants are presented with single numbers presented aurally, and must add each number they hear to the previous number and click the correct sum on the screen.
Period: Overall Study
Arm/Group | Cognitive Training Plus Treatment as Usual | Treatment as Usual (TAU)
Started | 24 | 22
Completed | 15 | 19
Not Completed | 9 | 3
Not completed — Lost to Follow-up | 4 | 2
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Participant reported exclusion criterion after study enrollment. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training Plus Treatment as Usual | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.75 (14.53) | 29.68 (10.28) | 31.80 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 22 | 20 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 21 | 39
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 24 | 22 | 46
Negative Urgency Scale-Short (subscale of Short UPPS-P Scale) [Mean (Standard Deviation); unit: units on a scale] — UPPS-P: Short Version of Urgency, (lack of) Premeditation, (lack of) Perseverance, Sensation Seeking, Positive Urgency scale.
  Negative Urgency Scale-Short: The range for this scale is 1-4, scored here such that higher scores reflect worse outcomes (higher levels of this type of impulsivity).
  units on a scale | 3.29 (0.41) | 3.28 (0.37) | 3.29 (0.39)
Positive Urgency Scale-Short (subscale of Short UPPS-P Scale) [Mean (Standard Deviation); unit: units on a scale] — UPPS-P: Short Version of Urgency, (lack of) Premeditation, (lack of) Perseverance, Sensation Seeking, Positive Urgency scale
  Positive Urgency Scale-Short: The range for this scale is 1-4, scored here such that higher scores reflect worse outcomes (higher levels of this type of impulsivity).
  units on a scale | 2.26 (0.72) | 2.47 (0.99) | 2.36 (0.85)
Stop-Signal Reaction Time (SSRT) [Mean (Standard Deviation); unit: milliseconds] — Population: Two participants in each arm did not complete the stop-signal task. In the cognitive training arm, 1 participant reported an exclusion criterion and discountined participation prior to completion of this task. 1 additional participant did not attend their session in which this task was to be completed.
  In the TAU arm, 1 participant dropped out of the study prior to completion of this measure, and 1 additional participant was not able to complete the task because of time constraints.
  milliseconds
    number analyzed (Participants) | 22 | 20 | 42
    (all) | 197.22 (99.73) | 216.22 (59.59) | 206.27 (82.66)

OUTCOME MEASURES:

1. Primary Outcome: Average Score on Negative Urgency Scale at Discharge
Description: This scale assesses tendencies towards impulsive action in response to negative emotion. The scale ranges from 1-4, with higher scores indicating more problems with this type of impulsivity.
Time Frame: Admission and at study completion (day of discharge), an average of two weeks. Scores reported below are at day of discharge.
Population: Note: two participants in the Treatment as Usual condition did not answer all questions for the Negative Urgency scale at discharge, so an average score was not computed, resulting in 17 participants with complete data.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Treatment as Usual: Participants in the Treatment As Usual group will receive usual treatment in the partial hospitalization program.
Arm/Group | Cognitive Training Plus Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 15 | 17
units on a scale | 3.17 (0.53) | 3.19 (0.30)
Statistical Analysis 1: Comparison: Cognitive Training Plus Treatment as Usual vs Treatment as Usual; A 2 (condition: TAU, TAU + cognitive training) x 2 (time) repeated-measures Analysis of Variance (ANOVA) was used to test change in negative urgency at time 1 (admission) and time 2 (discharge), and whether participants differ in their average change in negative urgency as a function of condition (interaction of condition X time; reported below); Test type: Superiority; p = 0.95, ANOVA; Repeated-measures ANOVA. P-value reflects the significance of the interaction term (condition x time)

2. Primary Outcome: Average Score on the Short Positive Urgency Scale at Discharge
Description: This scale assesses tendencies towards impulsive action in response to positive emotion. The scale ranges from 1-4, with higher scores indicating more problems with this type of impulsivity.
Time Frame: Admission and at study completion (day of discharge), an average of two weeks. Scores reported below are at discharge.
Population: Note: one participant in the Treatment as Usual condition did not answer all questions for the Positive Urgency scale at discharge, so an average score was not computed, resulting in 18 participants with complete data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training Plus Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 15 | 18
units on a scale | 2.07 (0.77) | 2.39 (0.81)
Statistical Analysis 1: Comparison: Cognitive Training Plus Treatment as Usual vs Treatment as Usual; A 2 (condition: TAU, TAU + cognitive training) x 2 (time) repeated-measures Analysis of Variance (ANOVA) was used to test change in positive urgency at time 1 (admission) and time 2 (discharge), and whether participants differ in their average change in positive urgency as a function of condition (interaction of condition X time; reported below); Test type: Superiority; p = 0.64, ANOVA; Repeated-measures ANOVA. P-value reflects the significance of the interaction term (condition x time)

3. Secondary Outcome: Estimated Stop-Signal Reaction Time (SSRT) on Stop-Signal Task (ms) at Discharge
Description: The SSRT (measured in ms) is the primary behavioral outcome measure of the Stop-Signal Response Inhibition task. It is an estimate of the average amount of time required to stop an action on this task.
Time Frame: Baseline and at study completion (discharge), an average of two weeks. Scores reported below are at discharge.
Population: 4 participants in the Cognitive Training plus Treatment as Usual group did not complete the Stop Signal task at discharge, for various reasons including: no-show to data collection session (1), equipment problem (1), clinical issues interfering with data collection (1), and time constraints (1); this resulted in a total of 11 participants with data for this task in this arm.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Cognitive Training Plus Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 11 | 19
milliseconds | 224.87 (50.61) | 236.69 (62.08)
Statistical Analysis 1: Comparison: Cognitive Training Plus Treatment as Usual vs Treatment as Usual; A 2 (condition: TAU, TAU + cognitive training) x 2 (time) repeated-measures Analysis of Variance (ANOVA) was used to test change in stop-signal reaction time at time 1 (admission) and time 2 (discharge), and whether participants differ in their average change in stop-signal reaction time as a function of condition (interaction of condition X time; reported below); Test type: Superiority; p = 0.91, ANOVA — Repeated-measures ANOVA. P-value reflects the significance of the interaction term (condition x time)

4. Secondary Outcome: Feasibility of Assessing Change in Event-related Potentials (ERPs) During a Stop-Signal Task in a Partial Hospital Population
Description: We evaluated the feasibility of using EEG to assess event-related potentials during the Stop-Signal task, in an acute partial hospital setting. This involves testing the percentage of participants who are able to complete and provide ERP data for the stop-signal task.
Time Frame: Baseline and at study completion (discharge), an average of two weeks. Baseline data and discharge data are shown separately below.
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Training Plus Treatment as Usual | Treatment as Usual
Number analyzed (Participants) | 24 | 22
Participants
  Baseline | 7 | 4
  Discharge | 5 | 2

5. Secondary Outcome: Completion Rates
Description: The percentage of participants enrolled in the cognitive training arm who complete the training sessions and the discharge session.
Time Frame: At study completion, an average of two weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Training Plus Treatment as Usual
Number analyzed (Participants) | 24
Participants | 15

6. Secondary Outcome: Average Perceived Helpfulness of Training
Description: This is a study-specific measure developed by the investigators to capture self-reported perceived helpfulness of the intervention. It consists of two separate questions that assess "how helpful" the Go/NoGo task and PASAT tasks were perceived to be. Each question is rated on a 1 ("completely disagree") to 7 ("completely agree") scale, with higher scores indicating better outcomes (i.e., greater perceived helpfulness of the task). Scores shown below are averages for each of these two items.
Time Frame: At study completion, an average of two weeks.
Population: One participant did not fill out this measure due to clinical issues interfering with data collection, resulting in 14 participants with available data. One additional participant filled out the measure but declined to fill out the item assessing perceived helpfulness of the PASAT, resulting in 13 participants available for anaylsis for this specific item.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training Plus Treatment as Usual
Number analyzed (Participants) | 14
units on a scale
  PASAT Perceived Helpfulness Rating: number analyzed (Participants) | 13
  PASAT Perceived Helpfulness Rating | 3.92 (1.44)
  Go/NoGo Perceived Helpfulness Rating | 5.07 (1.69)

7. Post Hoc Outcome: Average Score on Distress Intolerance Index (DII) Scale at Discharge
Description: This scale assesses self-reported difficulties tolerating distress. Total scores range from 0 to 40, with higher scores indicating greater difficulties tolerating distress.
Time Frame: as for outcome 1
Population: Note: two participants in the Cognitive Training plus Treatment as Usual arm, and 3 participants in the Treatment as Usual arm, did not answer all questions for the Distress Intolerance Index at discharge, so an average score was not computed, resulting in smaller sample sizes for these analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training Plus Treatment as Usual | Treatment as Usual (TAU)
Number analyzed (Participants) | 13 | 16
units on a scale | 21.77 (10.17) | 22.75 (9.21)
Statistical Analysis 1: Comparison: Cognitive Training Plus Treatment as Usual vs Treatment as Usual (TAU); A 2 (condition: TAU, TAU + cognitive training) x 2 (time) repeated-measures Analysis of Variance (ANOVA) was used to test change in distress intolerance at time 1 (admission) and time 2 (discharge), and whether participants differ in their average change in distress intolerance as a function of condition (interaction of condition X time; reported below); Test type: Superiority; p = .24, ANOVA; Repeated-measures ANOVA. P-value reflects the significance of the interaction term (condition x time)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the duration of a participant's study participation (approximately two weeks, corresponding to the overall length of partial hospitalization).
Arm/Group | Cognitive Training Plus Treatment as Usual | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 0/24 | 0/22

LIMITATIONS AND CAVEATS:
Recruitment for this trial was terminated early, prior to reaching the target sample size, due to the recruitment site shutting down during the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT03527550/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT03527550/SAP_001.pdf